CLINICAL TRIAL: NCT02649985
Title: Microglial Activation PET Brain Imaging in Multiple Sclerosis, Alzheimer's Disease, and Other Neurological and Neuropsychiatric Diseases
Brief Title: PET Brain Imaging in Multiple Sclerosis, Alzheimer's Disease, and Other Neurological and Neuropsychiatric Diseases
Acronym: MAPET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, TARUN SINGHAL, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P002329
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Alzheimer's Disease
MeSH Terms: conditions — Multiple Sclerosis; Alzheimer Disease | interventions — 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Relapsing-Remitting Multiple Sclerosis (Experimental): Subjects meeting the definition for RRMS by the International Panel Criteria, who are active, as defined by at least one MS relapse in the past 12 months, at least one gadolinium enhancing lesion on a MRI within 12 months of enrollment, or at least one new FLAIR bright lesion on MRI within 6 months of enrollment.
  The study will be performed in two phases. In the early pilot phase, 8 subjects with multiple sclerosis will undergo both [C-11]PBR28 PET scan and [F-18]PBR06 PET scan. At the end of this phase, a formal interim analysis will be performed and if imaging characteristics of [F-18]PBR06 are found non-inferior to or better than [C-11]PBR28, the rest of the study will be completed using [F-18]PBR06. On the other hand, if [F-18]PBR06 is found to be inferior to [C-11]PBR28, the rest of the study will be pursued using [C-11]PBR28.
  Interventions: Drug: [F-18]PBR06; Drug: [C-11]PBR28
- Progressive Multiple Sclerosis (Experimental): Subjects meeting the definition for SPMS/PPMS (Primary Progressive Multiple Sclerosis) by International Panel Criteria and who have demonstrated deterioration in EDSS score in last 1 year.
  Interventions: Drug: [F-18]PBR06
- Alzheimer's Disease (Experimental): Subjects meeting the definition for probable AD based on NINDS-ADRDA criteria. In terms of severity of disease, the investigators will select subjects with mild AD, as defined by Mini-Mental Status Examination (MMSE) score of 20-26.
  Interventions: Drug: [F-18]PBR06
- Healthy Control (Experimental): This group will serve as non disease population.
  Interventions: Drug: [F-18]PBR06
- Multiple Sclerosis Ocrelizumab (Experimental): Subjects who have already been prescribed Ocrelizumab by their treating MS neurologist, but have not yet started the first Ocrelizumab infusion.
  Subjects will undergo two separate visits for [F-18]PBR06 PET scans, once before starting Ocrelizumab and the second visit 3 months after completion of the initial Ocrelizumab doses.
  Interventions: Drug: [F-18]PBR06
- Multiple Sclerosis Foralumab (Experimental): Subjects will undergo 3 separate visits for [F-18]PBR06 PET scans, once before initiating treatment with Foralumab, the second visit 3 months after starting Foralumab, and the third visit 6 months after starting Foralumab.
  Interventions: Drug: [F-18]PBR06
- Multiple Sclerosis Steroids Treatment (Experimental): Subjects who have already been prescribed steroids by their treating MS neurologist, but have not yet initiated treatment.
  Subjects will undergo two separate visits for [F-18]PBR06 PET scans: one before steroid treatment and one after steroid treatment.
  Interventions: Drug: [F-18]PBR06

INTERVENTIONS:
Drug: [F-18]PBR06 — PET radiopharmaceutical
  Other Names: [F-18] PBR06
Drug: [C-11]PBR28 — PET radiopharmaceutical
  Other Names: [C-11] PBR28
  Arms: Relapsing-Remitting Multiple Sclerosis

SUMMARY:
The specific aims of the study are:

Primary: To determine the presence and regional distribution of microglial activation, as assessed by Fluorine-18 (18F) labeled "Peripheral Benzodiazepine Receptor 06" (PBR06) -PET, in subjects with active Relapsing Remitting Multiple Sclerosis (RRMS), Secondary Progressive Multiple Sclerosis (SPMS), and Alzheimer's Disease (AD) as compared to healthy controls

Secondary:

1. To assess the relationship between microglial activation and clinical variables including disease severity and comorbidities (such as pain, fatigue and/or depression), as well as clinical MRI findings (such as lesions and atrophy)
2. A pilot substudy aims to establish the non-inferiority of [F-18]PBR06 as compared with Carbon-11 [C-11] labeled "Peripheral Benzodiazepine Receptor 28" (PBR28) PET in patients with RRMS.

Hypothesis: The working hypothesis is that there is microglial activation in multiple sclerosis and Alzheimer's disease as compared to healthy controls and that the pattern/ regional distribution of microglial activation is different in Multiple Sclerosis (MS) versus AD and correlates with disease severity and comorbidities.

In addition, the investigators hypothesize that [F-18]PBR06-PET scans will be at least as good as [C-11]PBR28-PET scans, the current gold standard.

DETAILED DESCRIPTION:
Four groups of subjects will be recruited:

1. Subjects meeting the definition for RRMS by the International Panel Criteria, who are active, as defined by at least one MS relapse in the past 12 months, or at least one gadolinium enhancing lesion on Magnetic Resonance Imaging (MRI) within 3 months of enrollment.
2. Subjects meeting the definition for SPMS by International Panel Criteria and who have demonstrated deterioration in Expanded Disability Status Scale (EDSS) score in last 1 year
3. Subjects meeting the definition for probable AD based on National Institute of Neurological and Communicable Diseases-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria. In terms of severity of disease, we will select subjects with mild AD, as defined by Mini-Mental Status Examination (MMSE) score of 20-26.
4. Healthy Controls

The study will be performed in two phases. In the early pilot phase, 8 subjects with RRMS will undergo both [C-11]PBR28 PET scan and [F-18]PBR06 PET scan. At the end of this phase, a formal interim analysis will be performed and if imaging characteristics of [F-18]PBR06 are found non-inferior to or better than [C-11]PBR28, rest of the study will be completed using [F-18]PBR06. All subjects will also undergo 3-Tesla (3T) MRI of the brain.

The goal sample size is 30 subjects including 6 healthy controls, 8 subjects with relapsing remitting MS, 8 subjects with secondary progressive MS (SPMS), and 8 subjects with AD.

Subjects will be recruited by the PI, one of the other co-investigators, or a staff member listed on the protocol at the Partners MS Center and the Behavioral Neurology Clinic of Brigham and Women's Hospital.

Side Effects Monitoring:

No side effects from the radiopharmaceuticals are expected. The dose of radiopharmaceutical being administered in this study is below that at which we would expect any effect, including physical dependence and addiction. Subjects will be exposed to a small amount of radiation. The radiotracer will be prepared in such a way as to ensure that it is sterile and pyrogen free, and its radiochemical purity (RCP) will be determined using Silica Gel-Instant Thin Layer Chromatography and/or high pressure liquid chromatography (HPLC). In addition, because both [F-18]PBR06 and [C-11]PBR28 are non-FDA approved radioligands, their use for this study will be reviewed by Radioactive Drugs Research Committee.

Subject Safety:

Subject monitoring during MRI and PET scans will be performed using a 2-way intercom system between the scanner operator and subject and by visual monitoring of the subject through the window into the scan room (the subject is visible to the operator at all times).

Subjects will need to lie still in the PET camera for period of 120 min, and subjects may find it uncomfortable to remain still over this time. Therefore, as mentioned above, subjects will be given the opportunity to take a break for up to 20 minutes after 70 minutes of PET scanning, following which the last 30 minutes of scanning will be completed. A standard head-support device will be used to make the subjects comfortable during the scanning.

If subjects find an intravenous catheter or duration of scanning too uncomfortable, they are free to withdraw from the study at any time.

The MRI scans take place in a confined space that makes some people claustrophobic. Claustrophobic individuals will be excluded from the study. Also during the scan the subject will hear loud banging noises and will therefore wear ear plugs to reduce this noise.

Recruitment Process:

Physicians at the Partners MS Center and the Brigham and Women's Hospital (BWH) Behavioral Neurology clinic may present the study to a subject during a regular scheduled clinic visit. If the subject is interested in the study, a copy of the consent form will be given. At the time of the subject's initial screening visit, a licensed physician investigator will answer any questions the subject may have regarding the study and subsequently obtain informed consent. In accordance with NIH guidelines, efforts will be made to attain a mix of study participants, in terms of gender and racial/ethnic representation.

Consent Process:

Informed consent will be obtained from the subjects by a licensed physician investigator on the study protocol. If the investigator is a clinician from the MS Center or Behavioral Neurology clinic, they will not be allowed to obtain consent from their own patients. Existing MS Center or Behavioral Neurology clinic subjects may be sent a letter describing the study and a copy of the consent document. Interested subjects are directed to contact research staff via a telephone number provided in the letter inviting participation in the study to set up a screening visit. They will have the opportunity to discuss the study with research study staff prior to giving consent as outlined above. Subjects approached for participation in the study during a routine clinical visit will have the opportunity to participate in the study at that time or they may choose to return for participation at another time in the future. All subjects will be informed that they are free to withdraw consent from the study at any time without affecting the quality or type of care that they receive at BWH. Subjects will be informed that they may not qualify for the study if their genetic analysis reveals that they are low affinity binders for translocator protein (TSPO).

Monitoring and Quality Assurance:

During the study period, subjects will be followed by their clinical neurologists for adverse events and disease progression. If problems are reported to their physicians, they will receive care as is normally performed. In addition, the Principal Investigator (PI) will review all laboratory results of tests undergone by the subjects during the study period and help co-ordinate any necessary care with patient's primary providers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 70 years. For Alzheimer's Disease patients and healthy controls, the age range is going to be 18 to 85 years. This is because Alzheimer's disease subjects are usually older and it'd be difficult to recruit Alzheimer's patients who are younger than 70 years. Multiple Sclerosis, on the other hand, is a disease of a younger population.
2. For RRMS, it needs to be active, which is defined as at least one relapse in the past 12 months, at least one gadolinium enhancing lesion on MRI within 12 months of enrollment or at least one new FLAIR bright lesion on MRI within 6 months of enrollment.
3. For SPMS, deterioration in EDSS score in the last year is required.
4. For the subjects in the Ocrelizumab arm, only the subjects who have already been prescribed Ocrelizumab by their treating MS neurologist but have not yet started the first infusion, will be included.
5. For the Foralumab arm, patients enrolled in approved IRB protocols (2021P000105, 2022P000005, 2022P001075) will be enrolled.
6. For the steroids arm, only subjects who have already been prescribed steroids by their treating MS neurologist, but have not yet initiated treatment, will be included.
7. AD subjects with MMSE score of 20-26.
8. Subjects willing to undergo PET and MRI imaging
9. Subjects willing and able to give informed consent

Exclusion Criteria:

1. Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
2. Individuals with bipolar disease and schizophrenia
3. Concurrent medical conditions that contraindicate study procedures.
4. Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
5. Claustrophobia
6. Non-MRI compatible implanted devices
7. For the Ocrelizumab arm, subjects already on Ocrelizumab will be excluded. 8. For the steroids arm, subjects who have already started steroid treatment will be excluded.

9. For the Ocrelizumab arm, steroids arm, and longitudinal arm, subjects with abnormal serum creatinine will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake values (SUV)/Standardized uptake value ratios (SUVR) | Baseline, 3 months, and 6 months
  PET imaging measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham MS Center, 60 Fenwood Road, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singhal T, Cicero S, Rissanen E, Ficke J, Kukreja P, Vaquerano S, Glanz B, Dubey S, Sticka W, Seaver K, Kijewski M, Callen AM, Chu R, Carter K, Silbersweig D, Chitnis T, Bakshi R, Weiner HL. Glial Activity Load on PET Reveals Persistent "Smoldering" Inflammation in MS Despite Disease-Modifying Treatment: 18 F-PBR06 Study. Clin Nucl Med. 2024 Jun 1;49(6):491-499. doi: 10.1097/RLU.0000000000005201. Epub 2024 Apr 17. PMID 38630948